CLINICAL TRIAL: NCT02231229
Title: Rapid Detection of Rifampin and Isoniazid Resistance by PCR Before Tuberculosis (TB) Treatment Initiation: a National Multicenter Randomized Clinical Trial
Brief Title: Rapid Detection of Rifampin and Isoniazid Resistance by PCR Before Tuberculosis (TB) Treatment Initiation
Acronym: FAST-TB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P120130 AOM12317; IDRCB2013-A01406-39 (Other: FRENCH AUTHORITY)
Record Dates: First submitted 2014-07-03; First posted 2014-09-04 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Tuberculosis
Keywords: Pulmonary tuberculosis; Mycobacterium tuberculosis (MTB); Drug Resistance (DR); Isoniazid (INH or H); Rifampicin (RIF or RMP or R); Pyrazinamide (PZA or Z); Ethambutol (EMB or E); Fast-TB; Isoniazid, Rifampicin, Pyrazinamide (HRZ); Isoniazid, Rifampicin, Pyrazinamide, Ethambutol (HRZE); drug susceptibility testing (DST); Acid-Fast Bacilli (AFB+); Polymerase Chain Reaction (PCR)
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Sclerotylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCR-based strategy (Experimental): PCR-based strategy: after testing for isoniazid and rifampin resistance using a molecular testing with PCR (GenoType ®MTB DR plus), patients will receive HRZ combination therapy (INH , RIF, PZA) if no resistance is detected
  Interventions: Other: PCR-based strategy
- conventional therapy (Active Comparator): Conventional therapy: based on the standard of care in France: initiation of the standard 4 drug regimen INH, RIF, PZA, and EMB, until drug susceptibility testing (DST) results are available.
  Interventions: Drug: conventional therapy

INTERVENTIONS:
Other: PCR-based strategy — Treatment based on the results of detection of resistance to isoniazid and rifampicin using PCR (GenoType ® Mycobacterium Tuberculosis Drug Resistance (MTBDR)plus 2.0) in a smear positive patient with pulmonary tuberculosis: initiation of a 3 drug combination (isoniazid (H / INH); rifampicin (R /RIF); pyrazinamide (Z / PZA)) if no resistance is detected and treatment based on suspected resistance in case of INH and/or RIF resistant strain.
  Other Names: HRZ combination therapy
  Arms: PCR-based strategy
Drug: conventional therapy — Initiation of a standard 4 drug combination (isoniazid (H / INH); rifampicin (R /RIF); pyrazinamide (Z / PZA); ethambutol (EMB or E)) until the results of DST are available.
  Other Names: 4 drug combination (HRZE)
  Arms: conventional therapy

SUMMARY:
French guidelines currently recommend to initiate a 4-drug containing regimen associating isoniazid (INH or H), rifampicin (RIFor RMP or R), pyrazinamide (PZA or Z) and ethambutol (EMB or E) pending the results of drug susceptibility testing (DST). The rationale behind routine use of EMB is to prevent the emergence of resistance to rifampicin (RMP), in case of primary resistance to INH. Hence, early detection of resistance to INH and RIF using molecular testing in Mycobacterium tuberculosis could allow early adaptation of antituberculosis treatment: i) start with a 3-drug containing regimen (i.e. INH, RIF, and PZA); ii) early enforcement of treatment when resistance is suspected, pending in depth susceptibility testings.

the duration of treatment is 6 months or 12 months.

DETAILED DESCRIPTION:
The impact of rapid detection of resistance with PCR has been poorly evaluated in low-endemic countries. In France, primary resistance to isoniazid and rifampicin were estimated at, respectively, 5.2%, and 1.2 %. Based on these estimates, French guidelines currently recommends to initiate a 4-drug containing regimen associating isoniazid (INH or H), rifampicin (RIFor RMP or R), pyrazinamide (PZA or Z) and ethambutol (EMB or E) pending the results of drug susceptibility testing (DST). The rationale behind routine use of EMB is to prevent the emergence of resistance to rifampicin (RMP), in case of primary resistance to INH. Hence, early detection of resistance to INH and RIF using molecular testing in Mycobacterium tuberculosis could allow early adaptation of antituberculosis treatment: i) start with a 3-drug containing regimen (i.e. INH, RIF, and PZA), in patients with fully susceptible isolates (currently 95% of cases); ii) early enforcement of treatment when resistance is suspected, pending in depth susceptibility testings. GenoType ®MTB DR plus sensitivity for RIF and INH resistance detection has been estimated at 100% and 83%, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* with active pulmonary tuberculosis (TB) and positive respiratory samples on microscopic examination for acid-fast bacilli (AFB+,) who are eligible for a standard TB treatment with a 4 drug combination
* PCR (Genotype MTBDR Plus v2.0, Hain Lifescience) result available within the first 7 days of tuberculosis treatment.
* who are seeking care in France (metropolitan or overseas) and accept a follow-up of 18 to 24 months after inclusion.
* who have had a prior clinical examination

Exclusion Criteria:

* Refusal to participate in the study
* Prior history of TB treatment
* For women of child bearing age, pregnancy, willing to become pregnant or breastfeeding
* Patient without healthcare insurance (French social security)
* Patient participating in another clinical trial
* Any condition that might compromise, in the investigator's opinion, patient's compliance with the protocol.
* Results of cultures available at enrollment
* No HIV testing available within the last 3 months prior to inclusion in the study.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with treatment success at the end of TB treatment | 6 or 12 months after enrollment
  TB treatment success (cure certain or probable cure) at the end of TB treatment
  * cure certain: negative sputum cultures or negative sputum direct examination in a patient who has completed treatment and have never filled the definition of treatment failure.
  * probable cure: clinical and radiological improvement of symptoms associated with tuberculosis in a patient who has completed treatment and have never filled the definition of treatment failure.
  * completed treatment: patients who took more than 80% of prescribed treatment.
  * clinical improvement: improvement in overall score of Teeter AND no weight loss
  * radiological improvement: between baseline and end of treatment
  * failure: if Positive sputum culture after 5 months of treatment, death during treatment whatever the cause, treatment interrupted for more than two months, decision of the clinician to change TB treatment because of the suspicion of failure after 5 months of TB treatment

SECONDARY OUTCOMES:
Proportion of patients with relapse | within 12 months after the end of TB treatment
  positive culture of respiratory sample after TB treatment and after having had negative cultures during treatment or decision by the clinician to restart treatment because of suspicion of relapse
Proportion of patients with failure | 6 or 12 months after enrollment
  proportion of patients with treatment changes or discontinuations including the proportion of subjects stopping strategy and treatment assigned at randomization, and the delay between the stop and inclusion.
  Will not be considered modifications or discontinuations:
  * adaptation of treatment on the results of susceptibility testing in the conventional arm (adaptations following the susceptibility in the PCR arm will therefore be considered as a modification).
  * switching to bitherapy in the 2 arms.
Capillary drug concentration, for each of the prescribed treatment in hair segments | at 2 and 6 months
  measure of drug concentrations in hair segments, for each of the prescribed treatment, in order to estimate treatment observance and if drug hair concentrations are associated with therapy success or toxicity
Incidence and nature of grade 3 or grade 4 adverse events related or not to TB treatments | 6 months or at the latest 12 months after enrollment
  comparison between the 2 arms of incidence and nature of grade 3 or grade 4 adverse events related or not to TB treatments
Direct medical costs associated with each strategy | within 18 or at the latest 12 months after enrolment
  comparison of direct medical costs induced by PCR strategy and by conventional strategy

CONTACTS AND LOCATIONS:
Overall Officials: Yazdan Yazdanpanah, MD-PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Bichat Claude Bernard Hospital, Paris
  - Bichat hospital, Paris

IPD SHARING:
Plan to Share IPD: Undecided